CLINICAL TRIAL: NCT03644329
Title: Effect of Resistance Training Variable Manipulation (Intensity and Volume) on Body Composition, Fatigability and Functional Capacity in Postmenopausal Breast Cancer Survivors.
Brief Title: Effect of Resistance Training Variable Manipulation in Postmenopausal Breast Cancer Survivors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Fábio Lera Orsatti, Principal Investigator, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE: 82691818.0.0000.5154
Record Dates: First submitted 2018-08-14; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer Survivors; Postmenopause
Keywords: Breast Cancer Survivors; resistance Training; fatigability; Body Composition; Functional capacity
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group, CT (Other): In the CT, the postmenopausal breast cancer survivers does not perform exercise.
  Interventions: Other: Control group
- Lower-load resistance training (LL) (Experimental): In the LL, the postmenopausal breast cancer survivers will be submitted to 12 weeks of resistance training with low loads ( i.e. three sets with 30% of one-repetition maximum).
  Interventions: Other: Lower-load resistance training (LL)
- Higher-load resistance training (HL) (Experimental): In the HL, the postmenopausal breast cancer survivers will be submitted to 12 weeks of resistance training with high loads (i.e. three sets with 80% of one maximum repetition).
  Interventions: Other: Higher-load resistance training (HL)
- Higher-volume resistance training (HV) (Experimental): In the HV, the postmenopause breast cancer survivers will be submitted to 12 weeks of resistance training with high volume ( i.e. six sets with 80% one maximum repetition).
  Interventions: Other: Higher-volume resistance training (HV)

INTERVENTIONS:
Other: Control group — The volunteers will not performed the interventions.
  Arms: Control group, CT
Other: Lower-load resistance training (LL) — The volunteers will be perform the resistance training, three times a week for 12 weeks on non-consecutive days, three sets with 30% of 1RM and repetition until or close to failure in each set and 1.5-min of rest between sets and exercises.
  Arms: Lower-load resistance training (LL)
Other: Higher-load resistance training (HL) — The volunteers will be perform the resistance training, three times a week for 12 weeks on non-consecutive days, three sets with 80% of 1RM and repetition until or close to failure in each set and 1.5-min of rest between sets and exercises.
  Arms: Higher-load resistance training (HL)
Other: Higher-volume resistance training (HV) — The volunteers will be perform the resistance training, three times a week for 12 weeks on non-consecutive days, six sets with 80% of 1RM and repetition until or close to failure in each set and 1.5-min of rest between sets and exercises.
  Arms: Higher-volume resistance training (HV)

SUMMARY:
This study intends to evaluate the impact of resistance training variable manipulation (intensity and volume) on body composition, fatigability and functional capacity in postmenopausal breast cancer survivors.

DETAILED DESCRIPTION:
The treatment for breast cancer (chemotherapy, radiotherapy and hormone therapy) provokes collateral effects,such as muscle mass and strength losses, increase of fat mass, fatigue and disability and reduced quality of life in postmenopausal breast cancer survivors. The resistance training is assumed as a non-pharmacologic interventions in postmenopausal breast cancer survivors. However, it is unclear whether the manipulation of training variables (intensity and volume) maximize the effects of resistance training on body composition, fatigability and functional capacity in postmenopausal breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal breast cancer survivors;
* No supervised or unsupervised exercise at least for six months prior to the study.

Exclusion Criteria:

* Alcoholics;
* No controlled blood pressure and glucose;
* Presence of myopathies, arthropathies, and neuropathies;
* Presence of muscle, thromboembolic and gastrointestinal disorders, infection diseases.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-13 (Actual); Primary Completion 2018-11-10 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation the Fatigability | pre and post intervention (i.e. 12 weeks)
  The fatigability will be evaluate by 60 maximum voluntary isometric contractions (3 s contraction, 2 s rest) in knee extensors at 70 degree

SECONDARY OUTCOMES:
Four- meter walk test | pre and post intervention (i.e. 12 weeks)
  The volunteers will walk 4 meter. The time will be computed to determine the gait velocity (m/s).
Fat mass | pre intervention and post intervention (i.e. 12 weeks)
  The fat mass (kg) will be assessed via dual-energy x-ray absorptiometry scanning (iDXA; GE Healthcare-Luna, Madison, WI; software Encore version 14.10).
Muscle strength | pre and post intervention (i.e. 12 weeks)
  Muscle strength will be evaluated by one repetition maximum (1RM) test.
Six Minutes-walk test (6MWT) | pre and post intervention (i.e. 12 weeks)
  The volunteers will walk 6 minutes. The distance (meters) will be recorded after completes the test. The 6MWT will be performed indoor, on a flat floor in a sports court.
Timed Up and Go test | pre and post intervention (i.e. 12 weeks)
  The volunteers will be advised to get up from a chair, walk three meters, turn around, go back to the chair, and sit down. The time (seconds) will be recorded. The test will be performed indoor, on a flat floor in a sports court.
Five-times-sit-to-stand test | pre and post intervention (i.e. 12 weeks)
  The volunteers will rise from a chair and returned to the seated position as quickly as possible for five repetitions. The time will be recorded (seconds).
Muscle mass | pre and post intervention (i.e. 12 weeks)
  The muscle mass (kg) will be assessed via dual-energy x-ray absorptiometry scanning (iDXA; GE Healthcare-Luna, Madison, WI; software Encore version 14.10).
10-meter walk test | pre and post intervention (i.e. 12 weeks)
  The volunteers will walk 10 meters. The gait speed will be evaluated (m/s). The test will be performed indoor, on a flat floor in a sports court.
400-meter walk test | pre and post intervention (i.e. 12 weeks)
  The volunteers will walk 400 meters. The gait speed will be evaluated (m/s). The test will be performed indoor, on a flat floor in a sports court.
900-meter walk test | pre and post intervention (i.e. 12 weeks)
  The volunteers will walk 900 meters. The gait speed will be evaluate (m/s). The test will be performed indoor, on a flat floor in a sports court.

OTHER OUTCOMES:
Rate of force development (RFD) | pre and post intervention (i.e. 12 weeks)
  RFD will be measured by a rapid maximum isometric voluntary contraction of the one-sidedly knee extension force pulses of right leg.
Electromyography | pre and post intervention (i.e. 12 weeks)
  Quadriceps electromyography
Physical activity level | pre and post intervention (i.e. 12 weeks)
  The International Physical Activity Questionnaire short form (IPAQ) will be used to measure the level (time spent) of physical activities during the day. The questionnaire records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. The level of physical activity will be quantified by the sum of the four levels of intensity.
Evaluation the quality of life | pre and post intervention (i.e. 12 weeks)
  The 36-Item Short Form Health Survey (SF-36) will be used to measure the overall quality of life aspects in the following domains: functional capacity, physical limitations, pain, overall health, vitality, social aspects, emotional limitations and mental health.
Self-report fatigue | pre and post intervention (i.e. 12 weeks)
  The Brief Fatigue Inventory will be used for measured the self-report fatigue.
Cytokines | pre and post intervention (i.e. 12 weeks)
  Blood samples (16 ml) will be collected between 7:30 AM and 9:00 AM after an overnight fast (10-12 hours). The blood samples (venous) will be collected by a dry tube with gel separator or EDTA (vacuum-sealed system; Vacutainer, England). The sample will be centrifuged for 10 minutes (3.000 rpm) and samples will be separated and stocked (-80 C) for futures analysis. The blood indicators will be measured (enzyme-linked immunosorbent assay method) with Touch equipment and R&D kits (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Fábio L Orsatti, PhD, Principal Investigator — Federal University of Triângulo Mineiro
Locations (1):
- Post-degree program in physical education, Uberaba, MG - Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes J, Powell-Griner E, Lethbridge-Cejku M, Heyman K. Aging differently: Physical limitations among adults aged 50 years and over: United States, 2001-2007. NCHS Data Brief. 2009 Jul;(20):1-8. No abstract available. PMID 19627658
- [Background] Martin LG, Freedman VA, Schoeni RF, Andreski PM. Trends in disability and related chronic conditions among people ages fifty to sixty-four. Health Aff (Millwood). 2010 Apr;29(4):725-31. doi: 10.1377/hlthaff.2008.0746. PMID 20368601
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] McGinn AP, Kaplan RC, Verghese J, Rosenbaum DM, Psaty BM, Baird AE, Lynch JK, Wolf PA, Kooperberg C, Larson JC, Wassertheil-Smoller S. Walking speed and risk of incident ischemic stroke among postmenopausal women. Stroke. 2008 Apr;39(4):1233-9. doi: 10.1161/STROKEAHA.107.500850. Epub 2008 Feb 21. PMID 18292379
- [Background] Freiberger E, de Vreede P, Schoene D, Rydwik E, Mueller V, Frandin K, Hopman-Rock M. Performance-based physical function in older community-dwelling persons: a systematic review of instruments. Age Ageing. 2012 Nov;41(6):712-21. doi: 10.1093/ageing/afs099. Epub 2012 Aug 10. PMID 22885845
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Lyons RA, Perry HM, Littlepage BN. Evidence for the validity of the Short-form 36 Questionnaire (SF-36) in an elderly population. Age Ageing. 1994 May;23(3):182-4. doi: 10.1093/ageing/23.3.182. PMID 8085500
- [Background] Nunes PRP, Oliveira AA, Martins FM, Souza AP, Orsatti FL. Effect of resistance training volume on walking speed performance in postmenopausal women: A randomized controlled trial. Exp Gerontol. 2017 Oct 15;97:80-88. doi: 10.1016/j.exger.2017.08.011. Epub 2017 Aug 10. PMID 28804047
- [Background] Straight CR, Brady AO, Evans E. Sex-specific relationships of physical activity, body composition, and muscle quality with lower-extremity physical function in older men and women. Menopause. 2015 Mar;22(3):297-303. doi: 10.1097/GME.0000000000000313. PMID 25137244
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Buchner DM, Larson EB, Wagner EH, Koepsell TD, de Lateur BJ. Evidence for a non-linear relationship between leg strength and gait speed. Age Ageing. 1996 Sep;25(5):386-91. doi: 10.1093/ageing/25.5.386. PMID 8921145
- [Background] Reid KF, Fielding RA. Skeletal muscle power: a critical determinant of physical functioning in older adults. Exerc Sport Sci Rev. 2012 Jan;40(1):4-12. doi: 10.1097/JES.0b013e31823b5f13. PMID 22016147
- [Background] Rantanen T, Guralnik JM, Ferrucci L, Penninx BW, Leveille S, Sipila S, Fried LP. Coimpairments as predictors of severe walking disability in older women. J Am Geriatr Soc. 2001 Jan;49(1):21-7. doi: 10.1046/j.1532-5415.2001.49005.x. PMID 11207838
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Tseng LA, Delmonico MJ, Visser M, Boudreau RM, Goodpaster BH, Schwartz AV, Simonsick EM, Satterfield S, Harris T, Newman AB. Body composition explains sex differential in physical performance among older adults. J Gerontol A Biol Sci Med Sci. 2014 Jan;69(1):93-100. doi: 10.1093/gerona/glt027. Epub 2013 May 16. PMID 23682159
- [Background] Fragala MS, Clark MH, Walsh SJ, Kleppinger A, Judge JO, Kuchel GA, Kenny AM. Gender differences in anthropometric predictors of physical performance in older adults. Gend Med. 2012 Dec;9(6):445-56. doi: 10.1016/j.genm.2012.10.004. Epub 2012 Nov 2. PMID 23123187
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Orsatti FL, Nahas EA, Maesta N, Nahas-Neto J, Burini RC. Plasma hormones, muscle mass and strength in resistance-trained postmenopausal women. Maturitas. 2008 Apr 20;59(4):394-404. doi: 10.1016/j.maturitas.2008.04.002. Epub 2008 May 21. PMID 18499368
- [Background] Lera Orsatti F, Nahas EA, Maesta N, Nahas Neto J, Lera Orsatti C, Vannucchi Portari G, Burini RC. Effects of resistance training frequency on body composition and metabolics and inflammatory markers in overweight postmenopausal women. J Sports Med Phys Fitness. 2014 Jun;54(3):317-25. PMID 24739294
- [Background] Orsatti FL, Nahas EA, Nahas-Neto J, Maesta N, Orsatti CL, Fernandes CE. Effects of resistance training and soy isoflavone on body composition in postmenopausal women. Obstet Gynecol Int. 2010;2010:156037. doi: 10.1155/2010/156037. Epub 2010 May 18. PMID 20490353
- [Background] Senechal M, Bouchard DR, Dionne IJ, Brochu M. The effects of lifestyle interventions in dynapenic-obese postmenopausal women. Menopause. 2012 Sep;19(9):1015-21. doi: 10.1097/gme.0b013e318248f50f. PMID 22473250
- [Background] Haddock BL, Wilkin LD. Resistance training volume and post exercise energy expenditure. Int J Sports Med. 2006 Feb;27(2):143-8. doi: 10.1055/s-2005-865601. PMID 16475061
- [Background] Thompson R. Preventing cancer: the role of food, nutrition and physical activity. J Fam Health Care. 2010;20(3):100-2. PMID 20695357
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Krishnan K, Bassett JK, MacInnis RJ, English DR, Hopper JL, McLean C, Giles GG, Baglietto L. Associations between weight in early adulthood, change in weight, and breast cancer risk in postmenopausal women. Cancer Epidemiol Biomarkers Prev. 2013 Aug;22(8):1409-16. doi: 10.1158/1055-9965.EPI-13-0136. Epub 2013 May 29. PMID 23720403
- [Background] Majed B, Moreau T, Senouci K, Salmon RJ, Fourquet A, Asselain B. Is obesity an independent prognosis factor in woman breast cancer? Breast Cancer Res Treat. 2008 Sep;111(2):329-42. doi: 10.1007/s10549-007-9785-3. Epub 2007 Oct 16. PMID 17939036
- [Background] Patterson RE, Cadmus LA, Emond JA, Pierce JP. Physical activity, diet, adiposity and female breast cancer prognosis: a review of the epidemiologic literature. Maturitas. 2010 May;66(1):5-15. doi: 10.1016/j.maturitas.2010.01.004. Epub 2010 Jan 25. PMID 20097494
- [Background] Stone P, Hardy J, Broadley K, Tookman AJ, Kurowska A, A'Hern R. Fatigue in advanced cancer: a prospective controlled cross-sectional study. Br J Cancer. 1999 Mar;79(9-10):1479-86. doi: 10.1038/sj.bjc.6690236. PMID 10188894
- [Background] Courneya KS. Exercise in cancer survivors: an overview of research. Med Sci Sports Exerc. 2003 Nov;35(11):1846-52. doi: 10.1249/01.MSS.0000093622.41587.B6. PMID 14600549
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Martins da Silva RC, Rezende LF. Assessment of impact of late postoperative physical functional disabilities on quality of life in breast cancer survivors. Tumori. 2014 Jan-Feb;100(1):87-90. doi: 10.1700/1430.15821. PMID 24675497
- [Background] Rietman JS, Geertzen JH, Hoekstra HJ, Baas P, Dolsma WV, de Vries J, Groothoff JW, Eisma WH, Dijkstra PU. Long term treatment related upper limb morbidity and quality of life after sentinel lymph node biopsy for stage I or II breast cancer. Eur J Surg Oncol. 2006 Mar;32(2):148-52. doi: 10.1016/j.ejso.2005.11.008. Epub 2006 Jan 4. PMID 16387467
- [Background] Goedendorp MM, Gielissen MF, Verhagen CA, Bleijenberg G. Development of fatigue in cancer survivors: a prospective follow-up study from diagnosis into the year after treatment. J Pain Symptom Manage. 2013 Feb;45(2):213-22. doi: 10.1016/j.jpainsymman.2012.02.009. Epub 2012 Aug 25. PMID 22926087
- [Background] Berger AM, Mooney K, Alvarez-Perez A, Breitbart WS, Carpenter KM, Cella D, Cleeland C, Dotan E, Eisenberger MA, Escalante CP, Jacobsen PB, Jankowski C, LeBlanc T, Ligibel JA, Loggers ET, Mandrell B, Murphy BA, Palesh O, Pirl WF, Plaxe SC, Riba MB, Rugo HS, Salvador C, Wagner LI, Wagner-Johnston ND, Zachariah FJ, Bergman MA, Smith C; National comprehensive cancer network. Cancer-Related Fatigue, Version 2.2015. J Natl Compr Canc Netw. 2015 Aug;13(8):1012-39. doi: 10.6004/jnccn.2015.0122. PMID 26285247
- [Background] Barsevick AM, Irwin MR, Hinds P, Miller A, Berger A, Jacobsen P, Ancoli-Israel S, Reeve BB, Mustian K, O'Mara A, Lai JS, Fisch M, Cella D; National Cancer Institute Clinical Trials Planning Meeting. Recommendations for high-priority research on cancer-related fatigue in children and adults. J Natl Cancer Inst. 2013 Oct 2;105(19):1432-40. doi: 10.1093/jnci/djt242. Epub 2013 Sep 18. PMID 24047960
- [Background] Steindorf K, Schmidt ME, Klassen O, Ulrich CM, Oelmann J, Habermann N, Beckhove P, Owen R, Debus J, Wiskemann J, Potthoff K. Randomized, controlled trial of resistance training in breast cancer patients receiving adjuvant radiotherapy: results on cancer-related fatigue and quality of life. Ann Oncol. 2014 Nov;25(11):2237-2243. doi: 10.1093/annonc/mdu374. Epub 2014 Aug 5. PMID 25096607
- [Background] Hagstrom AD, Marshall PW, Lonsdale C, Cheema BS, Fiatarone Singh MA, Green S. Resistance training improves fatigue and quality of life in previously sedentary breast cancer survivors: a randomised controlled trial. Eur J Cancer Care (Engl). 2016 Sep;25(5):784-94. doi: 10.1111/ecc.12422. Epub 2015 Nov 23. PMID 26593858
- [Background] Serra MC, Ryan AS, Ortmeyer HK, Addison O, Goldberg AP. Resistance training reduces inflammation and fatigue and improves physical function in older breast cancer survivors. Menopause. 2018 Feb;25(2):211-216. doi: 10.1097/GME.0000000000000969. PMID 28832427
- [Background] Buffart LM, Ros WJ, Chinapaw MJ, Brug J, Knol DL, Korstjens I, van Weert E, Mesters I, van den Borne B, Hoekstra-Weebers JE, May AM. Mediators of physical exercise for improvement in cancer survivors' quality of life. Psychooncology. 2014 Mar;23(3):330-8. doi: 10.1002/pon.3428. Epub 2013 Oct 14. PMID 24123482
- [Background] Kalter J, Kampshoff CS, Chinapaw MJ, VAN Mechelen W, Galindo-Garre F, Schep G, Verdonck-DE Leeuw IM, Brug J, Buffart LM. Mediators of Exercise Effects on HRQoL in Cancer Survivors after Chemotherapy. Med Sci Sports Exerc. 2016 Oct;48(10):1859-65. doi: 10.1249/MSS.0000000000000976. PMID 27128668
- [Background] Hunter SK. Performance Fatigability: Mechanisms and Task Specificity. Cold Spring Harb Perspect Med. 2018 Jul 2;8(7):a029728. doi: 10.1101/cshperspect.a029728. PMID 28507192
- [Background] Enoka RM, Duchateau J. Translating Fatigue to Human Performance. Med Sci Sports Exerc. 2016 Nov;48(11):2228-2238. doi: 10.1249/MSS.0000000000000929. PMID 27015386
- [Background] Enoka RM, Baudry S, Rudroff T, Farina D, Klass M, Duchateau J. Unraveling the neurophysiology of muscle fatigue. J Electromyogr Kinesiol. 2011 Apr;21(2):208-19. doi: 10.1016/j.jelekin.2010.10.006. Epub 2010 Nov 10. PMID 21071242
- [Background] Enoka RM, Duchateau J. Muscle fatigue: what, why and how it influences muscle function. J Physiol. 2008 Jan 1;586(1):11-23. doi: 10.1113/jphysiol.2007.139477. Epub 2007 Aug 16. PMID 17702815
- [Background] Hunter SK, Pereira HM, Keenan KG. The aging neuromuscular system and motor performance. J Appl Physiol (1985). 2016 Oct 1;121(4):982-995. doi: 10.1152/japplphysiol.00475.2016. Epub 2016 Aug 11. PMID 27516536
- [Background] Poole DC, Burnley M, Vanhatalo A, Rossiter HB, Jones AM. Critical Power: An Important Fatigue Threshold in Exercise Physiology. Med Sci Sports Exerc. 2016 Nov;48(11):2320-2334. doi: 10.1249/MSS.0000000000000939. PMID 27031742
- [Background] Burnley M, Jones AM. Power-duration relationship: Physiology, fatigue, and the limits of human performance. Eur J Sport Sci. 2018 Feb;18(1):1-12. doi: 10.1080/17461391.2016.1249524. Epub 2016 Nov 3. PMID 27806677
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Marsh AP, Miller ME, Saikin AM, Rejeski WJ, Hu N, Lauretani F, Bandinelli S, Guralnik JM, Ferrucci L. Lower extremity strength and power are associated with 400-meter walk time in older adults: The InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1186-93. doi: 10.1093/gerona/61.11.1186. PMID 17167161
- [Background] Maffiuletti NA, Aagaard P, Blazevich AJ, Folland J, Tillin N, Duchateau J. Rate of force development: physiological and methodological considerations. Eur J Appl Physiol. 2016 Jun;116(6):1091-116. doi: 10.1007/s00421-016-3346-6. Epub 2016 Mar 3. PMID 26941023
- [Background] Fink J, Kikuchi N, Yoshida S, Terada K, Nakazato K. Impact of high versus low fixed loads and non-linear training loads on muscle hypertrophy, strength and force development. Springerplus. 2016 May 20;5(1):698. doi: 10.1186/s40064-016-2333-z. eCollection 2016. PMID 27350928
- [Background] Gurjao AL, Gobbi LT, Carneiro NH, Goncalves R, Ferreira de Moura R, Cyrino ES, Altimari LR, Gobbi S. Effect of strength training on rate of force development in older women. Res Q Exerc Sport. 2012 Jun;83(2):268-75. doi: 10.1080/02701367.2012.10599857. PMID 22808712
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] Burnley M. Estimation of critical torque using intermittent isometric maximal voluntary contractions of the quadriceps in humans. J Appl Physiol (1985). 2009 Mar;106(3):975-83. doi: 10.1152/japplphysiol.91474.2008. Epub 2009 Jan 15. PMID 19150854
- [Background] Klass M, Baudry S, Duchateau J. Voluntary activation during maximal contraction with advancing age: a brief review. Eur J Appl Physiol. 2007 Jul;100(5):543-51. doi: 10.1007/s00421-006-0205-x. Epub 2006 Jun 9. PMID 16763836
- [Background] Strasser B, Steindorf K, Wiskemann J, Ulrich CM. Impact of resistance training in cancer survivors: a meta-analysis. Med Sci Sports Exerc. 2013 Nov;45(11):2080-90. doi: 10.1249/MSS.0b013e31829a3b63. PMID 23669878